CLINICAL TRIAL: NCT05641129
Title: Acute PresentatiOn of CoLorectaL Cancer: an internatiOnal Snapshot-An International, Multi-centre Study of Emergency Presentations of Colorectal Cancer
Brief Title: Acute PresentatiOn of CoLorectaL Cancer: an internatiOnal Snapshot
Acronym: APOLLO
Status: Completed | Type: Observational
Sponsor: European Student Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: APOLLO Study
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal surgery; colorectal cancer; colonic stenting; emergency surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: Consecutive adult patients (≥18 years of age) presenting acutely (i.e. unplanned and non-elective presentation to hospital for urgent or emergency reasons) for symptoms of known or unknown colorectal cancer assessed by hospital surgical teams. Patients should be included regardless of operative or non-operative management, and curative or palliative intent.

SUMMARY:
APOLLO (Acute PresentatiOn of CoLorectaL Cancer: an internatiOnal snapshot) is an international, multi-centre, prospective observational study which will address this need and aims to describe the operative and non-operative management of emergency presentations of colon and rectal cancer in an international cohort.

DETAILED DESCRIPTION:
Primary aim: Describe the variation in the operative and non-operative management of emergency presentations of colon and rectal cancer in an international cohort.

Secondary aims:

* Identify risk factors for mortality (intraoperatively, at 30-days and at 90-days) and ostomy rates (at 30- and 90-days) in patients deemed for active management (i.e., not for palliative management) to develop a risk prediction model
* Validate risk criteria of large bowel obstruction in patients with previously known colorectal cancer undergoing neoadjuvant chemotherapy or awaiting elective surgery

Who?

* Patients aged 18 years and above presenting to the hospital acutely with colorectal cancer (CRC) for malignant large bowel obstruction (LBO), perforation, CRC-related haemorrhage or other reasons within the data collection periods. Both those managed with and without surgery will be included
* Patients with localised and metastatic disease will be included
* Patients with known colorectal cancer diagnoses will be included if they present acutely (e.g., with disease progression)
* Patients presenting acutely for the side effects of chemotherapy/radiotherapy of known cancers will be excluded

What? Data will be collected on patients' presenting status and symptoms, patient management strategies, and intraoperative and postoperative outcomes.

When? Prospectively over 2023 in consecutive 6-week data collection blocks between January and June with 90-day follow-up till September.

ELIGIBILITY:
Inclusion Criteria:

* Patient pathology: Patients admitted to the hospital acutely with primary colon AND/OR rectal adenocarcinoma and referred to general/colorectal surgical departments:
* Patients who are operated on for curative/palliative treatment of colorectal cancer
* Patients who are referred to general surgery for assessment (irrespective of if they proceed to surgery)
* New diagnoses of colorectal cancer
* Extent of cancer: All patients including extra-abdominal metastatic, intra-abdominal metastatic and non-metastatic disease
* Known cancer: Patients presenting for the first time with colorectal cancer AND/OR known colorectal cancer diagnosis with progression of disease. i.e. obstruction of known colorectal cancer
* Patient presentation: Symptomatic presentation of colorectal cancer i.e. large bowel obstruction, haemorrhage, perforation

Exclusion Criteria:

* Presenting for side effects of cancer treatment
* Patients with secondary cancers
* Previously included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (≥18 years of age) presenting acutely (i.e. unplanned and non-elective presentation to hospital for urgent or emergency reasons) for symptoms of known or unknown colorectal cancer assessed by hospital surgical teams. Patients should be included regardless of operative or non-operative management, and curative or palliative intent.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 90-day
  Mortality since day of presentation

SECONDARY OUTCOMES:
Secondary outcome 1 | 30-day
  Inpatient mortality, mortality since day of presentation
Secondary outcome 2 | 30- and 90-day
  Operative mortality rates
Secondary outcome 3 | 30- and 90-day
  Rates of primary anastomosis
Secondary outcome 4 | 30- and 90-day
  Stoma formation and reversal rates
Secondary outcome 5 | 90-day
  Rate and grade of surgical complications
Secondary outcome 6 | 30- and 90-day
  Rates of stenting in those with left-sided LBO, rates of stenting in those treated with palliative intent, rate of colonic stenting complications
Secondary outcome 7 | 30- and 90-day
  Rate of representation for patients managed nonoperatively
Secondary outcome8 | 30- and 90-day
  Rates of radiological assessment on admission
Secondary outcome 9 | 30- and 90-day
  Proportion of patients presenting acutely with large bowel obstruction with known colorectal cancer who had high risk criteria for obstruction (as defined by the FOXTroT obstruction criteria) at index assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Centre-summaries will be made available to respective centres for audit purposes.

REFERENCES:
- [Derived] EuroSurg Collaborative and STARSurg Collaborative. Global Use and Outcomes of Endoscopic Stenting in Acute Malignant Left-Sided Colonic Obstruction: A Secondary Analysis of APOLLO, An International, Prospective Cohort Study. Dis Colon Rectum. 2025 Dec 1;68(12):1458-1467. doi: 10.1097/DCR.0000000000003960. Epub 2025 Oct 10. PMID 41070782